CLINICAL TRIAL: NCT02744599
Title: Feasibility Trial for Detecting Drug-induced Respiratory Depression and Prompting for Self-rescue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Lara Brewer, Research Assistant Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB_00056695; R43NR015955 (NIH)
Record Dates: First submitted 2016-04-07; First posted 2016-04-20 (Estimated); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Healthy
Keywords: Feasibility trial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Device prompting (Experimental)
  Interventions: Device: Prompting breaths via recorded voice, vibrating massager, and/or muscle tetany
- Control (No Intervention): Patients receive standard of care

INTERVENTIONS:
Device: Prompting breaths via recorded voice, vibrating massager, and/or muscle tetany — Prompt volunteer to breathe using device to play recorded voice, massage the body, and/or apply muscle tetany
  Arms: Device prompting

SUMMARY:
This is a small trial to test feasibility of an idea for a potential device. The investigators tested the feasibility of prompting a volunteer to breathe when their breathing had slowed down during administration of anesthetic drugs.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesia (ASA) Class I and Class II male and female (non-pregnant/non-lactating) volunteers.
* Normal healthy individual as indicated by medical history and a physical examination.
* At least 18 years of age and less than 55 years of age.
* Negative drug screen.
* Uncomplicated airway anatomy.
* A Body Mass Index between 18 and 32.
* Are fully informed of the risks of entering the study and willingly provide written consent to enter the trial.
* Female subjects of child bearing potential will have a negative urine pregnancy test on the day the study is conducted.

Exclusion Criteria:

* Known or suspected neurological pathologies.
* A history of significant alcohol or drug abuse, a history of allergy to opioids or propofol, or a history of chronic drug requirement or medical illness that is known to alter the pharmacokinetics or pharmacodynamics of remifentanil and propofol.
* Known obstructive sleep apnea.
* Known or suspected hypersensitivity to any compound present in the study.
* Any potential subject suffering from medical problems that, in the judgment of the investigator, presents unacceptable risk to the volunteer are not eligible for enrollment.
* Vulnerable subject groups such as prisoners and the mentally disabled that are traditionally excluded from medical research are also excluded.
* The potential subject has taken any medication within 2 days prior to chosen drug administration, with the exception of oral contraceptives.
* The potential subject is wearing artificial nails.
* A positive urine pregnancy test (females only)
* Female subjects who are currently lactating & breast-feeding.
* A positive drug-screening test.
* The subject consumed food or fluids within 8 hours prior to start of each chosen drug administration.
* Any medications or alcohol within 2 days prior to start of the chosen drug administration, with the exception of oral contraceptives.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2013-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Breath prompting successful rate | Change in respiratory rate from baseline to the period 10 seconds after the breath prompt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Farney RJ, Johnson KB, Ermer SC, Orr JA, Egan TD, Morris AH, Brewer LM. Quantified Ataxic Breathing Can Detect Opioid-Induced Respiratory Depression Earlier in Normal Volunteers Infused with Remifentanil. Anesth Analg. 2025 Sep 1;141(3):507-515. doi: 10.1213/ANE.0000000000007124. Epub 2024 Aug 23. PMID 39178322
- [Derived] Ermer SC, Farney RJ, Johnson KB, Orr JA, Egan TD, Brewer LM. An Automated Algorithm Incorporating Poincare Analysis Can Quantify the Severity of Opioid-Induced Ataxic Breathing. Anesth Analg. 2020 May;130(5):1147-1156. doi: 10.1213/ANE.0000000000004498. PMID 32287122
- [Derived] Ermer S, Brewer L, Orr J, Egan TD, Johnson K. Comparison of 7 Different Sensors for Detecting Low Respiratory Rates Using a Single Breath Detection Algorithm in Nonintubated, Sedated Volunteers. Anesth Analg. 2019 Aug;129(2):399-408. doi: 10.1213/ANE.0000000000003793. PMID 30234539